CLINICAL TRIAL: NCT00772655
Title: Multicenter European Pilot Study of 90Yttrium-Ibritumomab Tiuxetan as First Line Therapy for Stage III - IV Follicular Lymphoma (and Selected Patients With Extended Stage II) Followed by Consolidation Rituximab for Patients in Complete Remission But With Persistent Molecular Disease
Brief Title: Zevalin® First Line in Follicular Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Christian Scholz M.D., PD Dr. med. Christian Scholz, Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT-No.:2006-005778-34; PEI-No.: 364/01; BFS-No.: 22461/2-2007-001
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Follicular Lymphoma
Keywords: Follicular Lymphoma; First line therapy; Zevalin; 90Yttrium-Ibritumomab Tiuxetan; Yttrium; Rituximab; Radio-immuno therapy
MeSH Terms: conditions — Lymphoma, Follicular | interventions — ibritumomab tiuxetan; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Therapy (Experimental): Induction therapy with a single course of 90Yttrium-Ibritumomab Tiuxetan (according to the standard procedure that includes Rituximab 250 mg/m2 plus 111Indium-Ibritumomab Tiuxetan for dosimetry on day one followed by Rituximab 250 mg/m2 and 90Y-Ibritumomab Tiuxetan 15 MBq/kg on day 8 or 9 up to a maximal dose of 12.000 MBq [if platelets are below 150000/µl only 11 MBq/kg are administered). Observation for patients achieving complete clinical and molecular response or partial clinical response. Consolidation/maintenance therapy with 4 weekly courses of Rituximab 375 mg/m2 followed by 4 bimonthly courses of Rituximab 375 mg/m2 for patients in clinical CR but with persistent Bcl-2 (t14;18)-positivity 6 months after 90Y-Ibritumomab Tiuxetan.
  Interventions: Drug: 90Yttrium-Ibritumomab Tiuxetan (Zevalin®)+Rituximab; Drug: Rituximab

INTERVENTIONS:
Drug: 90Yttrium-Ibritumomab Tiuxetan (Zevalin®)+Rituximab — A single course of 90Y-Ibritumomab Tiuxetan (according to the standard procedure that includes Rituximab 250 mg/m2 plus 111In-Ibritumomab Tiuxetan for dosimetry on day one followed by Rituximab 250 mg/m2 and 90Y-Ibritumomab Tiuxetan 15 MBq/kg on day 8 or 9 [if platelets are below 150000/µl only 11 MBq/kg are administered).
  Other Names: Zevalin®; Mabthera®
Drug: Rituximab — Consolidation/maintenance therapy with 4 weekly courses of Rituximab 375 mg/m2 followed by 4 bimonthly courses of Rituximab 375 mg/m2 for patients in clinical CR but with persistent Bcl-2-positivity 6 months after 90Y-Ibritumomab Tiuxetan.
  Other Names: Mabthera®

SUMMARY:
This is a European multicenter study of 90Yttrium-Ibritumomab Tiuxetan (90Y-Ibritumomab Tiuxetan) (Zevalin®) as a front line therapy for patients with follicular lymphoma grade I-IIIa and stage III-IV (as well as for selected patients with extended abdominal stage II). For patients with complete clinical remission but persistent molecular disease subsequent to 90Y-Ibritumomab Tiuxetan treatment a consolidation immunotherapy with Rituximab is added, to eradicate minimal residual disease.

DETAILED DESCRIPTION:
Only patients requiring treatment (B-symptoms, lymphoma progression > 50% within an observation period of 6 months or less, organ compression by lymphoma or bulky disease as defined by lesions above 5 cm on one axis) may enter the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 50 years old
* Follicular lymphoma grade I, II, or IIIa according to REAL/WHO classification
* Ann Arbor stage III, or IV, or stage II with disseminated abdominal disease requiring extensive abdominal irradiation
* No prior chemotherapy, immunotherapy, or irradiation. Furthermore, when receiving therapy as part of this "Zevalin® first line in follicular lymphoma" trial and up to six months after therapy has ended, patients may not participate in another clinical trial. If patients receive consolidation therapy with Rituximab, the six months period is counted from the end of the consolidation therapy.
* Lymphoma cells positive for CD20
* Measurable disease (two perpendicular diameters by either physical or radiological examination)
* WHO/ECOG performance status 0 - 2
* Written informed consent

Exclusion Criteria:

* Bone marrow involvement only
* Bone marrow infiltration > 25%
* Leukocytopenia < 2.500 /µl
* Thrombocytopenia < 100.000 /µl
* Bulk lesions > 10 cm
* CNS lymphoma manifestation
* Circulating tumor cells > 500 /µl
* Extensive pleural effusion/ascites (> 1000 ml as estimated by ultrasound/CT)
* Severe concomitant diseases (e.g. congestive heart failure, myocardial infarction within 6 months of study, severe uncontrolled hypertension, renal insufficiency requiring hemodialysis, pulmonary disease, liver disease)
* Abnormal liver function: transaminases or total bilirubin > 2 x upper limit of normal (ULN) (unless caused by the lymphoma)
* Abnormal renal function: serum creatinine > 2 x upper limit of normal (unless caused by the lymphoma)
* Previous malignancy other than non-melanoma skin cancer
* Pregnant or breast feeding female patients (negative pregnancy test required for women of fertile age), no effective contraception
* HIV positivity
* Known hypersensitivity to foreign proteins, murine antibodies, presence of human anti-murine antibodies (HAMA) reactivity
* Severe psychiatric illness

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-06 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Clinical and molecular remission rate after primary therapy with 90Y-Ibritumomab Tiuxetan | 6 months from entry onto trial

SECONDARY OUTCOMES:
Time to progression after treatment with 90Y-Ibritumomab Tiuxetan | 5 years from entry onto trial
Ability of consolidation therapy with Rituximab to induce molecular remission for CR patients not achieving molecular remission within 6 months after 90Y-Ibritumomab Tiuxetan | 5 years from entry onto trial
Safety and tolerability of 90Y-Ibritumomab Tiuxetan with particular respect to further therapy strategies in relapsed patients | 5 years from entry onto trial

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pezzutto, Prof., Principal Investigator — Dept. of Hematology, Charité Berlin, Germany; Christian Scholz, PD, Study Director — Dept. of Hematology, Charité Berlin, Germany

REFERENCES:
- [Derived] Rieger K, De Filippi R, Linden O, Viardot A, Hess G, Lerch K, Neumeister P, Stroux A, Peuker CA, Pezzutto A, Pinto A, Keller U, Scholz CW. 90-yttrium-ibritumomab tiuxetan as first-line treatment for follicular lymphoma: updated efficacy and safety results at an extended median follow-up of 9.6 years. Ann Hematol. 2022 Apr;101(4):781-788. doi: 10.1007/s00277-022-04781-3. Epub 2022 Feb 12. PMID 35150296
- [Derived] Scholz CW, Pinto A, Linkesch W, Linden O, Viardot A, Keller U, Hess G, Lastoria S, Lerch K, Frigeri F, Arcamone M, Stroux A, Frericks B, Pott C, Pezzutto A. (90)Yttrium-ibritumomab-tiuxetan as first-line treatment for follicular lymphoma: 30 months of follow-up data from an international multicenter phase II clinical trial. J Clin Oncol. 2013 Jan 20;31(3):308-13. doi: 10.1200/JCO.2011.41.1553. Epub 2012 Dec 10. PMID 23233718